CLINICAL TRIAL: NCT07177066
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of EDG-15400 in Healthy Adults
Brief Title: A Study of EDG-15400 in Healthy Adults
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Edgewise Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Basic Science
Other Study IDs: EDG-15400-101
Record Dates: First submitted 2025-08-27; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Healthy Adults

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A: Healthy Adult (Ages ≥18 to <60 years) Single Ascending Dose (Experimental): Single oral ascending dose in fasted healthy adults
  Interventions: Drug: EDG-15400; Drug: Placebo
- Part B: Healthy Adult (Ages ≥18 to <60 years) Multiple Ascending Doses (Experimental): Multiple oral ascending doses once daily in fasted healthy adults
  Interventions: Drug: EDG-15400; Drug: Placebo
- Part C: Healthy Adult (Ages ≥18 to <60 years) Food Effect and Relative Bioavailability (Experimental): Crossover food effect (fed versus fasted) single oral dose in healthy adults and relative bioavailability of liquid versus solid formulation
  Interventions: Drug: EDG-15400

INTERVENTIONS:
Drug: EDG-15400 — EDG-15400 is administered orally
Drug: Placebo — Placebo is administered orally
  Arms: Part A: Healthy Adult (Ages ≥18 to <60 years) Single Ascending Dose; Part B: Healthy Adult (Ages ≥18 to <60 years) Multiple Ascending Doses

SUMMARY:
The purposes of this Phase 1 study of EDG-15400 are to:

1. Learn about the safety of EDG-15400 after single and multiple doses in healthy adults
2. Learn about how EDG-15400 is tolerated after single and multiples doses in healthy adults
3. Evaluate the amount of EDG-15400 in the blood and urine after single and multiple doses in healthy adults
4. Evaluate the effect of a meal on the amount of EDG-15400 that is in the blood in healthy adults
5. Evaluate whether the amount of EDG-15400 in the blood is similar for the suspension and tablet forms of EDG-15400 in healthy adults

Participants will receive a single or multiple doses of EDG-15400 or a placebo by mouth.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give informed consent and follow all study procedures and requirements.
2. Healthy male or nonpregnant female, ages ≥18 to <60 years.
3. Body mass index (BMI) ≥18.5 to <35 kg/m2; weight ≥55 kg at Screening.
4. Absence of important health problems and essentially normal physical examination, normal laboratory screening tests, and normal electrocardiogram (ECG) with QTc interval corrected for heart rate using the Fridericia method (QTcF) ≤450 ms.

Exclusion Criteria:

1. Evidence of clinically significant abnormalities or disease.
2. Unless permitted by protocol, use of any prescription medication ≤ 4 weeks or investigational medication ≤ 12 weeks or ≤ 5 half-lives (whichever is longer) of dosing. Use of any non-prescription medication or herbal/nutritional supplement ≤ 5 days prior to dosing.
3. Donation or loss of > 1 unit (450 mL) of blood ≤ 1 month prior to dosing.
4. Females: nursing, lactating, or pregnant.
5. Females: breast implants.
6. Use of nicotine-containing products in the last 6 months prior to dosing.
7. History of substance abuse or dependency or history of recreational drug use within the last 2 years.
8. Alcohol consumption > 14 drinks per week for males (7 for females) within 45 days of screening.
9. Positive screen for drugs of abuse or alcohol or nicotine exposure test at Screening or Admission.

Additional protocol defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-08-20 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Safety: incidence of treatment-emergent adverse events | Up to 25 days of monitoring
  To determine the safety and tolerability of EDG-15400 when administered as single and multiple ascending doses to healthy adults

SECONDARY OUTCOMES:
Determination of Tmax | Up to 25 days
  Time to maximum concentration (Tmax)
Determination of Cmax | Up to 25 days
  Maximum observed concentration (Cmax)
Determination of AUC | Up to 25 days
  Area under the concentration-time curve (AUC)
Determination of t1/2 | Up to 25 days
  Elimination half-life (t1/2)
Determination of V/F | Up to 25 days
  Apparent volume of distribution after oral administration (V/F)
Determination of CL/F | Up to 25 days
  Apparent clearance of drug after oral administration (CL/F)
Determination of CLr | Up to 25 days
  Renal clearance (CLr)

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Inc., Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No